CLINICAL TRIAL: NCT04415151
Title: Investigation of Tofacitinib to Mitigate the Impact of COVID-19 (I-TOMIC) in Moderate SARS-CoV-2 (MODERATE I-TOMIC)
Brief Title: Tofacitinib for Treatment of Moderate COVID-19
Acronym: I-TOMIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to lack of enrollment reflecting the decrease in number of COVID infections. There were no safety and/or efficacy concerns involved in the decision to stop enrollment.
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Hyung Chun, Associate Professor of Internal Medicine, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000027848
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tofacitinib (Experimental): Tofacitinib will be administered in a dose of 10 mg PO BID until return to their clinical baseline (as defined by supplementary oxygen requirement), and then will continue to be administered at 5 mg PO BID for a total treatment duration of 14 days.
  Interventions: Drug: Tofacitinib 10 mg
- Placebo (Placebo Comparator): Matching placebo will be administered.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tofacitinib 10 mg — Tofacitinib will be administered in a dose of 10 mg twice daily by mouth (PO BID) until return to their clinical baseline (as defined by supplementary oxygen requirement), and then will continue to be administered at 5 mg PO BID for a total treatment duration of 14 days.
  Arms: Tofacitinib
Drug: Placebo — Matching placebo tablets will be administered.
  Arms: Placebo

SUMMARY:
The purpose of this randomized, double blinded, placebo controlled study is to assess the efficacy and safety of tofacitinib in hospitalized adult (18-99 years old) patients with SARS-CoV-2 and pneumonia who require supplemental oxygen and have serologic markers of inflammation but do not need mechanical ventilation.

DETAILED DESCRIPTION:
The purpose of this randomized, double blinded, placebo controlled Phase 2b study is to assess the efficacy and safety of tofacitinib in hospitalized adult (18-99 years old) male and female patients with SARS-CoV-2 and pneumonia who require supplemental oxygen and have serologic markers of inflammation but do not need mechanical ventilation (see Inclusion criteria). Sixty patients will be recruited to receive tofacitinib or placebo in addition to standard of care (SOC) in a 1:1 ratio.

Subjects will be screened during hospitalization. Patients with confirmed SARS-CoV-2 infection, and meeting all other Inclusion and Exclusion criteria, will be randomized to either treatment with tofacitinib or placebo in addition to SOC during hospitalization (dose adjusted, if required), with the exception of pre-specified immunomodulatory agents (as documented in the inclusion/exclusion criteria). Tofacitinib will be administered in a dose of 10 mg PO BID until return to their clinical baseline (as defined by need for supplementary oxygen), and will continue to be administered at 5 mg PO BID for a total duration of therapy of 14 days; follow-up off tofacitinib will continue up to Day 90. We anticipate completion of subject recruitment in 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
2. Participants with laboratory-confirmed novel coronavirus (SARS-CoV-2) infection as determined by polymerase chain reaction (PCR) or other commercially available or public health assay prior to Day 1.
3. Participants with evidence of pneumonia assessed by radiographic imaging (chest x ray or chest CT scan) AND Requiring ≥ 3L O2 OR ≥ 2L O2 and hsCRP > 70 mg/L
4. Participants who are hospitalized and receiving supportive care for COVID-19.
5. Participant (or legally authorized representative/surrogate) capable of giving signed informed consent.

Exclusion Criteria:

Medical Conditions:

1. Require mechanical ventilation or ECMO on Day 1 at the time of randomization.
2. Have current, or history of, venous thromboembolism (deep vein thrombosis or pulmonary embolism).
3. Have a personal or first-degree family history of blood clotting disorders.
4. Participants who are immunocompromised, with known immunodeficiencies, or taking potent immunosuppressive agents (eg, azathioprine, cyclosporine).
5. Participants with any current malignancy or lymphoproliferative disorders that requires active treatment
6. Females of child bearing potential who are pregnant or breastfeeding
7. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk associated with study participation or, in the investigator's judgment, make the participant inappropriate for the study.
8. Anticipated survival < 72 hours as assessed by the Investigator.

Infection History:

• Suspected or known active systemic bacterial, fungal, or viral infections (with the exception of COVID-19) including but not limited to:

* Secondary bacterial pneumonia;
* Active herpes zoster infection;
* Known active tuberculosis or history of inadequately treated tuberculosis;
* Known HBV, HCV, or HIV.

Prior/Concomitant Therapy:

Have received any of the following treatment regimens specified in the timeframes outlined below:

Within 4 weeks prior to the first dose of study intervention:

* Prior treatment with any JAK inhibitors, potent immunosuppressants, or any biologic agents including IL-6 inhibitors (eg, tocilizumab) or IL-1 inhibitors (eg, anakinra);
* Prior treatment with any potent cytochrome P450 inducer, such as rifampin, within the past 28 days or 5 half-lives, whichever is longer.

Within 48 hours prior to the first dose of study intervention:

o Treatment with herbal supplements.

Received >/= 20 mg/day of prednisone or equivalent for >/=14 consecutive days in the 4 weeks prior to screening.

Diagnostic Assessments:

* Severe hepatic impairment, defined as Child-Pugh class C.
* Severe anemia (hemoglobin <8 g/dL).
* ANY of the following abnormalities in clinical laboratory tests at screening, confirmed by a single repeat, if deemed necessary:
* WBC <1000/mm3
* Absolute lymphocyte count <500 cells/mm3;
* Absolute neutrophil count <1000 cells/mm3.
* Alanine transaminase/aspartate transaminase (ALT/AST) > 5 times the upper limit of normal;
* Estimated glomerular filtration rate (eGFR) < 40 mL/min/1.73 m2);

Other Exclusions:

* Known allergy to tofacitinib.
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Chun, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Health System, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tofacitinib | Placebo
Started | 13 | 11
Day 1 | 13 | 11
Day 2 | 13 | 9
Day 3 | 13 | 9
Day 4 | 12 | 9
Day 5 | 12 | 8
Day 6 | 11 | 8
Day 7 | 11 | 8
Day 8 | 9 | 5
Day 9 | 6 | 5
Day 10 | 5 | 5
Day 11 | 5 | 4
Day 12 | 5 | 4
Day 13 | 4 | 4
Day 14 | 3 | 4
Completed | 11 | 10
Not Completed | 2 | 1
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo group
- Tofacitinib: Tofacitinib group
- Total: Total of all reporting groups
Arm/Group | Placebo | Tofacitinib | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Disease Severity
Description: The primary objective of this study is to determine whether tofacitinib improves the clinical outcomes of patients with moderate SARS-CoV-2 infection as determined by the primary outcome measure: Proportion of subjects alive and not needing any form of mechanical ventilation, high flow oxygen, or ECMO by day 14.
Time Frame: 14 days
Population: All participants randomized and receiving at least 1 dose.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants taking Placebo with Usual Care.
- Tofacitinib: Participants taking Tofacitinib with Usual Care.
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 11 | 13
Participants | 5 | 10

2. Secondary Outcome: Clinical Improvement (Last Measure)
Description: Clinical improvement as measured by NIAID 8-point ordinal scale (i.e., 1 = death and 8 = Not hospitalized, no limitations on activities) at day 14.
  The scale is as follows:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities.
  Updated at the time of results entry, presented are the last clinical status for participants in the study (high scores are better outcomes).
Time Frame: Up to 14 days
Population: All participants randomized and receiving at least 1 dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 11 | 13
Participants
  Death | 1 | 1
  Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) | 0 | 1
  Hospitalized, on non-invasive ventilation or high flow oxygen devices | 2 | 0
  Hospitalized, requiring supplemental oxygen | 3 | 1
  Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (CovID19/otherwise) | 0 | 0
  Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care | 0 | 1
  Not hospitalized, limitation on activities and/or requiring home oxygen | 5 | 9
  Not hospitalized, no limitations on activities | 0 | 0

3. Secondary Outcome: Clinical Improvement (Improved Score)
Description: Clinical improvement as measured by NIAID 8-point ordinal scale (i.e., 1 = death and 8 = Not hospitalized, no limitations on activities) (days 3 through day 14):
  The scale is as follows:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities.
  Added at the time of results entry: this outcome presents those that improved at least 2 or more levels on the clinical scale (high scores are better outcomes).
Time Frame: Up to 14 days
Population: All participants randomized and receiving at least 1 dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 11 | 13
Participants | 5 | 9

4. Secondary Outcome: Time to Recovery
Description: Time to recovery [ Time Frame: Day 1 through Day 14] (Day of recovery is defined as the first day on which the subject satisfies one of the following three categories from the ordinal scale:
  1. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  2. Not hospitalized, limitation on activities and/or requiring home oxygen
  3. Not hospitalized, no limitations on activities)
Time Frame: Up to 14 days
Population: Of those that "recovered" within 14 days.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 5 | 10
days | 5.0 [3.0 to 8.0] | 5.0 [0.0 to 12]

5. Secondary Outcome: Time to Clinical Improvement
Description: Time to clinical improvement (defined as a 2-point increase on the NIAID 8-point ordinal scale (i.e., 1 = death and 8 = Not hospitalized, no limitations on activities).
  The scale is as follows:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities.
  Updated at the time of results entry, the follow up time frame was adjusted.
Time Frame: Up to 14 days
Population: Participants successfully follow up with.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 5 | 10
days | 5 [3 to 8] | 5 [0 to 10]

6. Secondary Outcome: Clinical Status
Description: Clinical status on the NIAID 8-point ordinal scale at day 30
  The scale is as follows:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities.
  Updated at the time of results entry, the follow up time frame was adjusted.
Time Frame: Up to 28 Days
Population: Participants (alive at end of 14 days) successfully followed up with.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 10 | 10
Participants
  Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) | 1 | 1
  Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (CovID19/etc) | 1 | 0
  Not hospitalized, limitation on activities and/or requiring home oxygen | 3 | 4
  Not hospitalized, no limitations on activities | 5 | 5

7. Secondary Outcome: Clinical Status
Description: Clinical status on the NIAID 8-point ordinal scale at day 60
  The scale is as follows:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities.
Time Frame: 60 Days
Population: Participants (alive at end of 14 days) successfully followed up with.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 8 | 10
Participants
  Hospitalized, on non-invasive ventilation or high flow oxygen devices | 1 | 1
  Not hospitalized, limitation on activities and/or requiring home oxygen | 4 | 1
  Not hospitalized, no limitations on activities | 3 | 8

8. Secondary Outcome: Clinical Status
Description: Clinical status on the NIAID 8-point ordinal scale at day 90
  The scale is as follows:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities.
Time Frame: 90 Days
Population: Participants (alive at end of 14 days) successfully followed up with.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 9 | 11
Participants
  Hospitalized, on non-invasive ventilation or high flow oxygen devices | 1 | 0
  Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (CovID19/etc) | 0 | 1
  Not hospitalized, limitation on activities and/or requiring home oxygen | 2 | 2
  Not hospitalized, no limitations on activities | 6 | 8

9. Secondary Outcome: Mortality
Description: Mortality rate at day 30 (28 Days- updated at time of results entry). Presented are a count of those participants that expired (all-cause) through the 28 day follow up. This outcome includes counts of those that expired during the study period (see adverse events All-Cause Mortality).
Time Frame: Up to 28 Days
Population: Participants successfully followed up with post study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 10 | 10
Participants | 1 | 1

10. Secondary Outcome: Mortality
Description: Mortality rate at day 60 (updated at time of results entry). Presented are a count of those participants that expired (all-cause) through the 60 day follow up. This outcome includes counts of those that expired during the study period (see adverse events All Cause Mortality).
Time Frame: 60 Days
Population: Participants successfully followed up with post study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 8 | 10
Participants | 1 | 1

11. Secondary Outcome: Mortality
Description: Mortality rate at day 90. Presented are a count of those participants that expired (all-cause) through the 90 day follow up. This outcome includes counts of those that expired during the study period (see adverse events All-Cause Mortality).
Time Frame: 90 Days
Population: Participants successfully followed up with post study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 9 | 11
Participants | 1 | 1

12. Secondary Outcome: Mechanical Ventilatory Support
Description: Proportion of patients requiring mechanical ventilatory support.
Time Frame: Up to 14 Days
Population: All participants randomized and receiving at least 1 dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 11 | 13
Participants | 1 | 2

13. Secondary Outcome: Mechanical Ventilatory Support Duration
Description: Duration of invasive mechanical ventilation (days).
Time Frame: Up to 14 Days
Population: Only those on invasive mechanical ventilation (days).
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 1 | 2
days | 2 [2 to 2] | 10.5 [10 to 11]

14. Secondary Outcome: Freedom From Mechanical Ventilation
Description: Invasive mechanical ventilation free days. The outcome was updated to present the number of participants that were without invasive mechanical ventilation while on study.
Time Frame: Up to 14 Days
Population: All participants randomized and receiving at least 1 dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 11 | 13
Participants | 10 | 11

15. Secondary Outcome: Additional Intervention
Description: Did the patient receive an intervention with additional immunomodulatory agent (i.e. IL-6 targeting therapy)? (y/n)
Time Frame: Up to 14 days
Population: All participants randomized and receiving at least 1 dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 11 | 13
Participants
  Yes | 0 | 0
  No | 11 | 13

16. Secondary Outcome: Viral Titer
Description: Change in SARS-CoV-2 viral titers during intervention. Upon entry of results, the time frame was updated to Day 7 to reflect the data collected in the terminated study. Nasopharyngeal (NP) swab were used and the visit window for Day 7 could include days between Day 5 to Day 9. Imputation for < LLOQ: N gene: "<200" is imputed to 2.0 log10 copies/mL (log10(200) - 0.3). ORF1ab gene: "<3000" is imputed to 3.2 log10 copies/mL (log10(3000) - 0.3). Missing Data were not imputed.
Time Frame: Day 7 (Day 5 to Day 9)
Population: All data collected on all participants
Measure: Mean (Standard Deviation); unit: log10 (copies/mL)
Arm/Group | Placebo | Tofacitinib
Number analyzed (Participants) | 7 | 8
log10 (copies/mL)
  SARS-CoV-2 Viral Load: N Gene BASELINE: number analyzed (Participants) | 7 | 7
  SARS-CoV-2 Viral Load: N Gene BASELINE | 3.30 (1.38) | 3.61 (1.07)
  SARS-CoV-2 Viral Load: N Gene 7 DAYS | 2.80 (1.00) | 2.50 (0.66)
  SARS-CoV-2 Viral Load: ORF1ab Gene BASELINE | 3.70 (0.79) | 3.92 (0.82)
  SARS-CoV-2 Viral Load: ORF1ab Gene 7 DAYS | 3.27 (0.25) | 3.24 (0.21)

17. Other Pre Specified Outcome: Adverse Events
Description: Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment. All adverse events are presented in the adverse event module.
Time Frame: Up to 14 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All Other Adverse Events and Serious Adverse Event data were collected up to 14 days, All Cause Mortality data were collected up to 90 days
Groups:
- Placebo: Participants received placebo and usual care.
- Tofacitinib: Participants received Tofacitinib and usual care.
Arm/Group | Placebo | Tofacitinib
All-Cause Mortality (participants affected / at risk) | 1/11 | 1/13
Serious Adverse Events (participants affected / at risk) | 2/11 | 2/13
Other Adverse Events (participants affected / at risk) | 10/11 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | Tofacitinib (N=13)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | Tofacitinib (N=13)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 7 (7)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 6 (6)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT04415151/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT04415151/SAP_001.pdf